CLINICAL TRIAL: NCT05764031
Title: Comparative Effects of Clinical Pilates Training and Aerobic Exercise on Menopausal Symptoms, Quality of Life, Sleep and Depression
Brief Title: Clinical Pilates and Aerobic Exercise in Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Serkan Usgu, Clinical Professor, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2020/114
Record Dates: First submitted 2023-03-01; First posted 2023-03-10 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Menopause
Keywords: Menopause; Aerobic exercise; Pilates; Depression; Sleep; Quality of life
MeSH Terms: conditions — Depression | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical pilates group (Experimental): The clinical pilates group received a total of 40 min of exercise training, including 5 min of warm-up exercises, 30 min of clinical pilates exercises and 5 min of cooldown exercises. Clinical Pilates training was performed as group sessions under the supervision of a physiotherapist Exercise training was provided to the clinical pilates group 2 days a week over a period of 8 weeks.
  Interventions: Other: Clinical pilates exercise
- Aerobic exercise group (Experimental): The aerobic exercise group received a total of 40 min of aerobic exercise training, including 5 min of warm-up exercises, 30 min of aerobic cycling exercise and 5 min of cooldown exercises. Aerobic exercises were performed individually under the supervision of a physiotherapist. Aerobic exercises were performed using an upright bike (HS-1200; Hattrick-Pro, Istanbul, Turkey). The exercises were planned as moderate-intensity exercises, at 60-70% of the maximum heart rate (MHR). Exercise training was provided to the aerobic exercise group 2 days a week over a period of 8 weeks.
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Other: Clinical pilates exercise — Clinical pilates is an exercise modality in which postural muscles are worked out with various body movements, and involves multi-muscle synergies that improve spinal stabilization, flexibility and endurance.
  Arms: Clinical pilates group
Other: Aerobic exercise — Aerobic exercise (also known as endurance activities, cardio or cardio-respiratory exercise) is physical exercise of low to high intensity that depends primarily on the aerobic energy-generating process.
  Arms: Aerobic exercise group

SUMMARY:
To the best of our knowledge, there is no study in the literature that examined the effects of clinical Pilates training on vasomotor symptoms, quality of life, depression, and sleep problems versus aerobic exercises in menopausal women. This study aimed to investigate the effects of clinical Pilates training and aerobic exercises on menopausal symptoms, depression and quality of life and sleep quality in menopausal women.

DETAILED DESCRIPTION:
Menopause is defined as the time in a woman's life when there is a decrease in ovarian function and permanent cessation of reproductive function. Identification of the healthcare needs of menopausal women requires special attention. During menopause, hormonal, physical and emotional changes occur as a result of decreased estrogen levels. Psychological, somatic and atrophic changes occur in the early stages of menopause and cardiovascular disease and osteoporosis during late menopause.

Due to the complex nature of menopause, various approaches are employed in the treatment of menopausal symptoms. Hormone Replacement Therapy (HRT) is one of them. However, prolonged use of combined estrogen/progesterone therapy may increase the risk of breast cancer. Among the conservative treatment methods, exercise is the most reliable and effective approach. Exercise provides similar benefits as HRT. The effects of exercise may vary with the initiation and type of exercise and the individual level of adherence to exercise. During exercise, cardiovascular, respiratory and musculoskeletal systems work together. In the short-term, regular exercise increases endurance, reduces stress and encourages better sleep patterns in a short period of time. In the longer term, exercise can reduce the risk of coronary artery disease (CAD), hypertension (HT) and type 2 diabetes.

Various exercise approaches are employed including aerobic exercise, yoga, pilates and relaxation exercises. Mixed findings on the outcomes of exercise have been reported in published studies. In a study examining the effects of aerobic exercise, yoga and diet on vasomotor symptoms (VMS) in menopausal women, exercise and diet were found to have no effect, whereas yoga showed beneficial effects on VMS. 12-week yoga and aerobic exercises were not effective in improving actigraphic sleep parameters in menopausal women with hot flashes. Contrastingly, a 6-week walking exercise program was demonstrated to improve sleep quality of postmenopausal women. A study evaluating the effects of aerobic exercise on estrogen level, fat mass and muscle mass versus resistance exercises in postmenopausal women found that resistance exercises were more effective in improving these parameters. Usgu et al. reported that 8-week aerobic walking exercises provided a reduction in somatic and psychological complaints, had no effect on urogenital symptoms but improved quality of life in premenopausal women. A meta-analysis of randomized trials aiming to determine the impact of low-to-moderate-intensity exercises on depressive symptoms in middle-aged and older women found that both types of exercises were effective in alleviating depressive symptoms. Moderate-intensity (VO2 max 60%) walking exercises practiced for 4 months showed greater effects on menopausal symptoms, physical activity, depression, satisfaction with life, self-esteem and feelings of loneliness compared to control.

On the other hand, Pilates is an exercise modality in which postural muscles are worked out with various body movements, and involves multi-muscle synergies that improve spinal stabilization, flexibility and endurance. The biopsychosocial effects of Pilates in menopausal women have been shown in many studies. Positive effects of a 12-week Pilates training on sleep quality, depression, fatigue and anxiety in postmenopausal women were previously demonstrated. An 8-week Pilates training was found to reduce depression by improving quality of life in menopausal women. A systematic review of published studies on the efficacy of Pilates exercises in the rehabilitation of several conditions including postmenopausal osteoporosis concluded that Pilates can be prescribed for effective management of postmenopausal osteoporosis. In a meta-analysis of the trials examining the effect of exercise on women with depression, Pilates training was shown to reduce depressive symptoms in postmenopausal women compared to control group in one study included in the analysis. In the same meta-analysis involving 25 studies, aerobic exercise training was found to provide similar effects on depressive symptoms when compared with other exercise methods.

To the best of our knowledge, there is no study in the literature that examined the effects of clinical Pilates training on vasomotor symptoms, quality of life, depression, and sleep problems versus aerobic exercises in menopausal women. This study aimed to investigate the effects of clinical Pilates training and aerobic exercises on menopausal symptoms, depression and quality of life and sleep quality in menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Womens between the ages of 40 and 65
* diagnosis of menopause by a gynecologist and willingness to participate in the study

Exclusion Criteria:

* Women with a systemic, cardiovascular or neurological disorder, surgical menopause, alcohol or substance abuse and those who missed more than 3 sessions of exercise training.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Menopause is defined as the time in a woman's life when there is a decrease in ovarian function and permanent cessation of reproductive function
Enrollment: 30 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Menopause Rating Scale | 8 weeks
  This self-report questionnaire consists of 11 items in 3 subscales including somatic, urogenital and psychological complaints. The somatic dimension measures joint and muscle problems, sleep disturbances, hot flashes and cardiac discomfort. The psychological domain measures physical and mental exhaustion, anxiety, irritability and depressive mood. The urogenital domain measures sexual problems, vaginal dryness/soreness and bladder. Each item is assigned a score between 0 and 4, and possible total scores range from 0 (asymptomatic) to 44 (highest degree of complaints). Domain scores range from 0 to 16 for the somatic and psychological domains and from 0 and 12 for the urogenital domain.

SECONDARY OUTCOMES:
36-Item Short Form Health Survey | 8 weeks
  The new short-form health survey (SF-36) was developed by Ware and Sherbourne. In this study, the Turkish version of the SF-36 questionnaire validated by Kocyigit was used for the assessment of quality of life. The tool consists of 36 items in eight sections, including physical functioning, physical role functioning, emotional role functioning, social role functioning, general health perceptions, bodily pain, vitality/energy and mental health. Each item is assigned a score between 0 and 100 and averaged to obtain the subscale scores.
Beck Depression Inventory | 8 weeks
  The Beck Depression Inventory was developed by Beck in 1961 for the measurement of the severity of depression. The scale consists of 21 items, including 2 items for emotions, 11 items for cognitions, 2 items for behaviors, 5 items for physical symptoms and 1 item for interpersonal symptoms. Each answer is scored between 0 and 3, with a possible total score ranging from 0 to 63. Higher scores denote more severe depressive symptoms.
Pittsburgh Sleep Quality Index | 8 weeks
  Pittsburgh Sleep Quality Index (PSQI) is composed of 24 questions. Among them, 19 questions are self-rated questions and 18 of them are scored. The latter 5 questions are responded by the bed partner or roommate. The tool consists of 7 components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each question is rated from 0 to 3. The sum of scores for the seven components yields the overall PSQI score. Higher scores indicate worse sleep quality

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Greendale GA, Lee NP, Arriola ER. The menopause. Lancet. 1999 Feb 13;353(9152):571-80. doi: 10.1016/S0140-6736(98)05352-5. PMID 10028999
- [Result] Santoro N, Epperson CN, Mathews SB. Menopausal Symptoms and Their Management. Endocrinol Metab Clin North Am. 2015 Sep;44(3):497-515. doi: 10.1016/j.ecl.2015.05.001. PMID 26316239
- [Result] Monteleone P, Mascagni G, Giannini A, Genazzani AR, Simoncini T. Symptoms of menopause - global prevalence, physiology and implications. Nat Rev Endocrinol. 2018 Apr;14(4):199-215. doi: 10.1038/nrendo.2017.180. Epub 2018 Feb 2. PMID 29393299
- [Result] Stojanovska L, Apostolopoulos V, Polman R, Borkoles E. To exercise, or, not to exercise, during menopause and beyond. Maturitas. 2014 Apr;77(4):318-23. doi: 10.1016/j.maturitas.2014.01.006. Epub 2014 Jan 24. PMID 24548848
- [Result] Hill DA, Crider M, Hill SR. Hormone Therapy and Other Treatments for Symptoms of Menopause. Am Fam Physician. 2016 Dec 1;94(11):884-889. PMID 27929271
- [Result] Reed SD, Guthrie KA, Newton KM, Anderson GL, Booth-LaForce C, Caan B, Carpenter JS, Cohen LS, Dunn AL, Ensrud KE, Freeman EW, Hunt JR, Joffe H, Larson JC, Learman LA, Rothenberg R, Seguin RA, Sherman KJ, Sternfeld BS, LaCroix AZ. Menopausal quality of life: RCT of yoga, exercise, and omega-3 supplements. Am J Obstet Gynecol. 2014 Mar;210(3):244.e1-11. doi: 10.1016/j.ajog.2013.11.016. Epub 2013 Nov 8. PMID 24215858
- [Result] Buchanan DT, Landis CA, Hohensee C, Guthrie KA, Otte JL, Paudel M, Anderson GL, Caan B, Freeman EW, Joffe H, LaCroix AZ, Newton KM, Reed SD, Ensrud KE. Effects of Yoga and Aerobic Exercise on Actigraphic Sleep Parameters in Menopausal Women with Hot Flashes. J Clin Sleep Med. 2017 Jan 15;13(1):11-18. doi: 10.5664/jcsm.6376. PMID 27707450
- [Result] Razzak ZA, Khan AA, Farooqui SI. Effect of aerobic and anaerobic exercise on estrogen level, fat mass, and muscle mass among postmenopausal osteoporotic females. Int J Health Sci (Qassim). 2019 Jul-Aug;13(4):10-16. PMID 31341450